CLINICAL TRIAL: NCT01864330
Title: Influence of Lachrymal Substitutes on Tear Film Thickness in Patients With Moderate Dry Eye Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: OPHT-28102012
Record Dates: First submitted 2013-05-03; First posted 2013-05-29 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Dry Eye Syndrome
Keywords: topical lubricants; optical coherence tomography; tear break up time; Schirmer I test
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dry Eye Syndrome I (Experimental): 20 patients with moderate dry eye syndrome
  Interventions: Device: Thealoz Duo®
- Dry Eye Syndrome II (Active Comparator): 20 patients with moderate dry eye syndrome
  Interventions: Device: Hyabak®
- Dry Eye Syndrome III (Active Comparator): 20 patients with moderate dry eye syndrome
  Interventions: Device: Hydrabak®

INTERVENTIONS:
Device: Thealoz Duo® — Eye Drops
  Arms: Dry Eye Syndrome I
Device: Hyabak® — Eye Drops
  Arms: Dry Eye Syndrome II
Device: Hydrabak® — Eye Drops
  Arms: Dry Eye Syndrome III

SUMMARY:
Dry eye syndrome is a highly prevalent ocular disease with an increasing incidence in the elderly population. Topically administered lubricants are the basis for treatment of this disease. However, information about the corneal residence time of topical lubricants is still sparse, therefore no ideal treatment regimen has been found.

Recently a new method for assessment of tear film thickness based on optical coherence tomography (OCT) has become available. The aim of the present study is to assess corneal residence time of three different formulations of topical lubricants, in particular Thealoz Duo® Eye Drops, Hyabak® Eye Drops and Hydrabak® Eye Drops in patients with moderate dry eye disease. In addition, standard tests for dry eye syndrome, such as the ocular surface disease index (OSDI©), Schirmer I test and determination of tear break up time (BUT) will be performed..

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* Signed and dated written informed consent.
* History of dry eye syndrome for at least 3 months
* Tear Break Up Time (BUT) ≤ 10 seconds or Schirmer I test ≤ 5 mm and ≥ 2mm
* OSDI (Ocular Surface Disease Index) ≤ 32 and ≥ 13
* Normal ophthalmic findings except dry eye syndrome, ametropia < 6 Dpt.
* No administration of topical lubricants 24 hours before the screening examination

Exclusion Criteria:

* Participation in a clinical trial in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition as judged by the clinical investigator
* Intake of parasympathomimetic or anti-psychotic drugs
* Wearing of contact lenses
* Glaucoma
* Treatment with corticosteroids in the 4 weeks preceding the study
* Topical treatment with any ophthalmic drug except topical lubricants in the 4 weeks preceding the study
* Ocular infection or clinically significant inflammation
* Ocular surgery in the 3 months preceding the study
* Sjögren's syndrome
* Stevens-Johnson syndrome
* History of allergic conjunctivitis
* Ametropia >= 6 Dpt
* Pregnancy, planned pregnancy or lactating
* Known hypersensitivity to any component of the study medication.
* Any medical or surgical history, disorder or disease such as acute or chronic severe organic disease
* Inability to understand the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Tear film thickness | Change in tear film thickness from predose to 10 ± 3 minutes, 20 ± 3 minutes, 40 ± 5 minutes, 60 ± 5 minutes, 120 ± 10 minutes and 240 ± 10 minutes after instillation
  Change in tear film thickness as measured with OCT.
  Total time frame is 4 hours

SECONDARY OUTCOMES:
Tear Break Up Time | change from screening to the last OCT measurement
  Total time frame is 14 days
Subjective evaluation of ocular comfort | change after instillation and after the last OCT measurement
  Ocular comfort will be assessed immediately after instillation and at the end of the study day.
  Total time frame is 4 hours.
Schirmer I test | change from screening to after the last OCT measurement
  Total time frame is 14 days
Visual Acuity | change from screening to after the last OCT measurement
  Total time frame is 14 days.
Intraocular Pressure | change from screening to after the last OCT measurement
  Total time frame is 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhoefer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Vienna, Austria